CLINICAL TRIAL: NCT00837707
Title: Aripiprazole for Pre-Existing Neuroleptic-Induced Tardive Dyskinesia: a Prospective 26-Week Observational Study
Brief Title: Aripiprazole for Neuroleptic-Induced Tardive Dyskinesia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taoyuan Psychiatric Center, Ministry of Health and Welfare, Executive Yuan, R.O.C. Taiwan (Other Government)
Collaborators: Department of Health (Ambiguous)
Responsible Party: Chia-Hsiang Chan/ Attending Psychiatrist of General Psychiatry, Taoyuan Mental Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMH-97-03
Record Dates: First submitted 2009-02-04; First posted 2009-02-05 (Estimated); Last update posted 2009-02-05 (Estimated); Status verified 2009-02

CONDITIONS: Dyskinesia, Drug-Induced
Keywords: aripiprazole; Tardive Dyskinesia
MeSH Terms: conditions — Dyskinesia, Drug-Induced; Tardive Dyskinesia | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: aripiprazole — Flexible dose: 5-30 mg/day
  Other Names: Abilify

SUMMARY:
The aim of the present study was to investigate the efficacy of aripiprazole in management of pre-existing neuroleptic-induced tardive dyskinesia

DETAILED DESCRIPTION:
Objective:A few case reports on the use of aripiprazole in neuroleptic-induced tardive dyskinesia have demonstrated positive effects. However its effectiveness in treatment of TD was still inconclusive. The aim of the present study was to investigate the efficacy of aripiprazole in management of pre-existing neuroleptic-induced tardive dyskinesia.

Method: Subjects with pre-existing neuroleptic-induced tardive dyskinesia were chosen from Taoyuan psychiatric center. Patients recruited would be treated with aripiprazole for cross-titration with previous antipsychotics in 8 weeks. We use AIMS, SAS, & BAS to assess the severity of TF and EPS. We record subjects' age, sex, and other factors which have influence at the treatment response. Subjects are assessed every two weeks in the first month and then monthly until six months.

ELIGIBILITY:
Inclusion Criteria:

* Female patients must agree to prevent from being pregnant during trial periods
* Meet psychotic disorder or mood disorder criteria of DSM-IV
* Patients must have psychiatric diseases that need to use antipsychotics for a long time
* They must meet DSM-IV research criteria for neuroleptics induce tardive dyskinesia
* No clinical significant major systemic diseases
* No special neurological diseases which would influence the assessment for EPS or TD
* Mentality is better than mild mental retardation
* Patients or .legal representatives agree to join in the research and sign informed consent.

Exclusion Criteria:

* Unstable major systemic diseases
* Had neurological disorder influenced to EPS assessment
* Substance abuse or dependence other then coffee or tobacco within 6 months before study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2008-06; Primary Completion 2009-08 (Estimated); Study Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
Total scores of AIMS | The change from baseline to study endpoint

SECONDARY OUTCOMES:
Total scores of PANSS | The change from baseline to study endpoint
Total scores of SAS | The change from baseline to study endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Hsiang Chan, M.D., Study Chair — Taoyuan Psychiatric Center, Ministry of Health and Welfare, Executive Yuan, R.O.C. Taiwan
Locations (1):
- Taoyuan Mental Hospital, Taoyuan District, Taiwan

REFERENCES:
- [Background] Aripiprazole improves neuroleptic-associated tardive dyskinesia, but it does not meliorate psychotic symptoms. Prog Neuropsychopharmacol Biol Psychiatry. 2008 Jul 1;32(5):1342-3. doi: 10.1016/j.pnpbp.2008.03.003. Epub 2008 Mar 18. No abstract available. PMID 18433967
- [Background] Lykouras L, Rizos E, Gournellis R. Aripiprazole in the treatment of tardive dyskinesia induced by other atypical antipsychotics. Prog Neuropsychopharmacol Biol Psychiatry. 2007 Oct 1;31(7):1535-6. doi: 10.1016/j.pnpbp.2007.06.010. Epub 2007 Jun 22. No abstract available. PMID 17614184
- [Background] Witschy JK, Winter AS. Improvement in tardive dyskinesia with aripiprazole use. Can J Psychiatry. 2005 Mar;50(3):188. doi: 10.1177/070674370505000321. No abstract available. PMID 15830835
- [Background] Grant MJ, Baldessarini RJ. Possible improvement of neuroleptic-associated tardive dyskinesia during treatment with aripiprazole. Ann Pharmacother. 2005 Nov;39(11):1953. doi: 10.1345/aph.1G255. Epub 2005 Oct 11. No abstract available. PMID 16219895